CLINICAL TRIAL: NCT00005735
Title: Controlling Asthma at School
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4944; R01HL068654 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-07

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To implement and evaluate a coordinated set of activities for asthma identification, education, management, and prevention in the predominantly minority inner city schools in the Detroit metropolitan area.

DETAILED DESCRIPTION:
BACKGROUND:

The study was part of an initiative "Interventions to Improve Asthma Management and Prevention at School". The Broad Agency Announcement was released in June, 1994.

DESIGN NARRATIVE:

The intervention was a combination of: targeted education for children with asthma, other children in the school, families, physicians and school personnel; concerted effort to change school policies working against effective self-management of asthma; community action/education to create awareness and support for the schools' efforts to control the disease. Open Airways for School, a proven educational program, was adapted for students in the Detroit metropolitan area as part of the intervention. This program was based on social cognitive theory while modeling effective asthma management behavior, involving students in activities where they mastered skills relevant to asthma management, and developing the students' sense of confidence to carry out asthma management tasks. For education of all students, a learning module called "Environmental Detective" was developed to complement the Michigan Model of comprehensive health education offered in classrooms in Michigan. The Environmental Detective game sensitized children without asthma to the problems of children with asthma. The intervention was evaluated through a controlled research design to determine if it had an impact on asthma morbidity, the number of days of limited activity of the child with asthma, and his or her academic performance.

The project was a collaboration of the University of Michigan School of Public Health and School of Medicine, the Henry Ford Hospital Center of Detroit, the Washtenaw County Health and Human Services Department, the American Lung Association of Michigan, and the State of Michigan Department of Education.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Clark — University of Michigan

REFERENCES:
- [Background] Clark NM, Brown R, Joseph CL, Anderson EW, Liu M, Valerio M, Gong M. Issues in identifying asthma and estimating prevalence in an urban school population. J Clin Epidemiol. 2002 Sep;55(9):870-81. doi: 10.1016/s0895-4356(02)00451-1. PMID 12393074
- [Background] Clark NM, Brown R, Joseph CL, Anderson EW, Liu M, Valerio MA. Effects of a comprehensive school-based asthma program on symptoms, parent management, grades, and absenteeism. Chest. 2004 May;125(5):1674-9. doi: 10.1378/chest.125.5.1674. PMID 15136375